CLINICAL TRIAL: NCT01608230
Title: Human Tumor Sequencing Project
Acronym: HuTS
Status: Completed | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Principal Investigator, Eric Topol, MD, Director, Scripps Translational Science Institute
Other Study IDs: 09-5270
Record Dates: First submitted 2012-05-25; First posted 2012-05-31 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is being done to learn more about genetic mutations in cancer cells and to find out how the development of new technologies can increase knowledge of these mutations and possibly predict an individual's response to certain treatments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a solid tumor or blood borne cancer
* 18 years or older
* Eligible to have blood drawn

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2010-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Determine biomarkers of clinical utility and copy number variants through genetic analysis. | four years

CONTACTS AND LOCATIONS:
Locations (1):
- Scripps Translational Science Institute, La Jolla, California, United States